CLINICAL TRIAL: NCT04247061
Title: Delivery of a Smoking Cessation Induction Intervention Via Virtual Reality (VR) Headset During a Dental Cleaning: Usability Study
Brief Title: Usability Study of a Smoking Cessation Intervention During a Dental Cleaning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 policies this usability pilot study was stopped after enrolling 4 participants.
Sponsor: Boston University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-39053; 1UG3DE028866 (NIH)
Record Dates: First submitted 2020-01-28; First posted 2020-01-29 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Smoking, Cessation
Keywords: Dental cleaning; Video; Text messages
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smoking Cessation intervention (Experimental): At a dental cleaning visit, participants will watch a brief educational video that provides guidance and advice on smoking cessation. Participants will then interact with a text program for a month to motivate them to use smoking cessation resources. Participants will also be required to make contact with the resources in order to demonstrate feasibility of study flow.
  Interventions: Other: Educational video; Other: Text-message program

INTERVENTIONS:
Other: Educational video — One of two different 10 minute educational videos on smoking cessation will be viewed by participants during a dental cleaning visit. The video that is watched will depend on participants' level of motivation to quit and project needs
Other: Text-message program — A one-month text message program to motivate and facilitate contact with smoking cessation resources.

SUMMARY:
The goal of this usability study is to pilot test the recruitment procedures, data acquisition methods, and text message program integration required to support the planning of a future clinical trial. Approximately 15 smokers who are patients of the Boston University Goldman School of Dental Medicine (BUGSDM) patient treatment center and have an upcoming dental prophylaxis or scaling and root planing (henceforth referred to as 'teeth cleaning') appointment will be recruited. During the dental cleaning, participants will watch a brief educational video that provides guidance and advice on smoking cessation.

At the end of the dental appointment, participants will complete a survey about their experience watching the video and their attitudes towards smoking cessation. Participants will also receive other smoking cessation resources with instructions on how to access the services. Participants will then use the one-month text message program developed by the investigators to motivate and facilitate contact with the smoking cessation resources.

At the end of the one-month text message program, participants will complete a survey about their experience during the text message program, their smoking habits, and attitudes towards smoking cessation. The duration of the study will be approximately six-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient of the Boston University, Henry M Goldman School of Dental Medicine patient treatment center
* Must have smoked 100 cigarettes or more (not e-cigarettes or vaping) in lifetime
* Must have smoked cigarettes (not e-cigarettes or vaping) 'most days' or 'every day' in the past week
* Must read and write fluently in English
* Must be willing to watch a video during the dental hygiene appointment
* Must have the visual capacity to watch a video
* Ability to wear in-ear headphones
* Must have a mobile phone capable of receiving and sending text messages (SMS)
* live in Greater Boston area for the next two months
* Have a cell phone carrier that can receive text message from our system

Exclusion Criteria:

-Planning to move out of the Greater Boston area within the next two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Borrelli, PhD, Principal Investigator — Henry M Goldman School of Dental Medicine
Locations (1):
- Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 subjects were enrolled (provided informed consent to participate). Of the 16 enrolled, 13 subjects completed the pre-dental visit activities (n=1 did not opt into the text message program, n=2 did not complete the baseline questionnaire) and were scheduled to attend the dental clinic visit.
Period: Overall Study
Arm/Group | Smoking Cessation Intervention
Started | 13 (13 Subjects completed the required pre-dental appointment study activities and were scheduled to attend the dental clinic)
Completed | 4
Not Completed | 9
Not completed — Could not attend dental clinic visit due to state mandated closure due to Covid-19 pandemic | 6
Not completed — Subjects canceled their dental hygiene appt. (& thus the research visit) due to Covid-19 concerns | 2
Not completed — Participant indicated inability to wear VR headset at dental appt. | 1

BASELINE CHARACTERISTICS:
Population: 16 subjects were enrolled (provided informed consent to participate)
Arm/Group | Smoking Cessation Intervention
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 7
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Smoking Cessation Education Program
Description: The number of participants who watched the video and used the text messaging for a month.
Time Frame: 6 weeks
Population: 16 participants provided informed consent. Of the 16, n=13 completed required pre-dental visit study activities and were scheduled to attend the clinic visit. Of the 13, n=4 completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Intervention
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Participant Acceptability Rate of the Program
Description: Participants were asked to rate the acceptability of the program by answering an investigator developed acceptability question with a scale of 1 to 7, where 1= the program was not acceptable and 7= the program was very acceptable. Scores could range from 1 to 7, and higher scores are associated with greater acceptability of the program.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale (1 to 7 scale)
Arm/Group | Smoking Cessation Intervention
Number analyzed (Participants) | 4
Units on a scale (1 to 7 scale) | 5.9 (1.3)

3. Primary Outcome: Participant Satisfaction With the Program
Description: Participants were asked to rate their satisfaction of the program by answering an investigator developed satisfaction question with a scale of 1 to 5, where 1= they were not satisfied with the program and 5= they were very satisfied with the program. Higher scores were associated with greater satisfaction with the program.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (1 to 5 scale)
Arm/Group | Smoking Cessation Intervention
Number analyzed (Participants) | 4
units on a scale (1 to 5 scale) | 4.5 (0.58)

4. Secondary Outcome: Attitudes About Smoking
Description: The number of subjects who 'agreed' or 'strongly agreed' that the educational video improved their attitude towards quitting smoking.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Intervention
Number analyzed (Participants) | 4
Participants | 4

5. Secondary Outcome: Change in Number of Cigarettes Smoked Per Day
Description: An investigator-developed survey will ask participants questions about the number of cigarettes smoked daily
Time Frame: Baseline, 6 weeks
Population: The change in the number of cigarettes smoked per day between baseline and follow-up cannot be computed because the one participant who reported smoking at follow-up did not report the number of cigarettes.
Arm/Group | Smoking Cessation Intervention
Number analyzed (Participants) | 0

6. Secondary Outcome: The Number of Participants With Quit Attempts Lasting ≥ 24 Hours
Description: The number of participants who attempted to quit smoking for 24 hours or more at follow-up because they wanted to quit (not due to hospitalization or illness) based on an investigator-developed survey that asked participants questions about the number of quit attempts lasting ≥ 24 hours
Time Frame: 6 weeks
Population: 16 participants provided informed consent. Of the 16, n=13 completed required pre-dental visit study activities and were scheduled to attend the clinic visit. Of the 13, 4 completed the study, however, quit attempts data were not collected from one participant, so there are only 3 participants for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Intervention
Number analyzed (Participants) | 3
Participants | 3

7. Secondary Outcome: Methods for Quitting Smoking
Description: An investigator-developed survey will ask participants questions about what methods they used to try to quit smoking
Time Frame: 6 weeks
Population: The number of participants who indicated that they used one or more methods to help them quit smoking (or help them make an attempt to quit smoking)
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Intervention
Number analyzed (Participants) | 3
Participants
  Acupuncture or hypnosis | 1
  Cold turkey (without aid) | 3
  Brochure or book | 1
  Gradually cutting back cigarettes | 2
  Nicotine replacement patch | 1
  Quit smoking mobile apps | 1
  Quit smoking text message program (other than VR study text message) | 2
  Quit smoking online program | 1
  Watched a video on how to stop smoking (other than video watched at dental visit) | 2

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Smoking Cessation Intervention
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Of the 16 enrolled subjects, n=13 completed required pre-dental visit activities & were scheduled to attend the clinic. Of the 13, n=4 completed the study (n=6 could not attend clinic due to Covid-19, state-mandated closure; n=2 canceled their dental appointment due to Covid-19 concerns; n=1 indicated inability to wear VR headset at the clinic). Thus, due to the Covid-19 pandemic restrictions, this usability study was terminated early leading to small numbers of subjects completing the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT04247061/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT04247061/SAP_002.pdf
  • Informed Consent Form (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT04247061/ICF_000.pdf